CLINICAL TRIAL: NCT05666141
Title: The Effect of Pharyngeal Electrical Stimulation (PES) on Peripheral Biomechanical Aspects of Deglutition
Brief Title: The Effect of Pharyngeal Electrical Stimulation on Peripheral Biomechanical Aspects of Deglutition
Acronym: PES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Phagenesis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: S65439
Record Dates: First submitted 2022-11-29; First posted 2022-12-27 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-05

CONDITIONS: Dysphagia Following Cerebrovascular Accident; Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (7):
- PES stimulation in volunteers (Experimental): 10 volunteers will receive PES stimulation. For healthy volunteers, the study protocol includes 1 stimulation trial. Each stimulation trial consists of 3 PES sessions. A session is a 10-minute stimulation, once per day. The sessions will be given on three consecutive days at optimal parameters, as reported by Fraser et al. (2003).
  Interventions: Device: Pharyngeal Electrical Stimulation
- Sham treatment in volunteers (Sham Comparator): 10 volunteers will receive Sham treatment. In the Sham condition, the same method and same device will be used. The time spent interacting with the patient will remain constant, including placement of the PES catheter which will be left in situ in the subject for the duration of intervention (10 minutes). However, the base-station will be set to 0 milliampere (mA), so Sham subjects do not receive any active electrical current.
  Interventions: Other: Sham treatment
- PES stimulation + PES stimulation in stroke patients (Experimental): Max 8 patients will receive PES stimulation twice. For patients, the protocol thus includes 2 stimulation trails. Each stimulation trial consists of 3 PES sessions, so they receive 6 PES sessions in total. A session is a 10-minute stimulation, once per day. The sessions will be given on three consecutive days at optimal parameters, as reported by Fraser et al. (2003).
  Interventions: Device: Pharyngeal Electrical Stimulation
- PES stimulation + Sham treatment in stroke patients (Other): Max 8 patients will receive PES stimulation and afterwards Sham treatment. During the first stimulation trial, they will receive 3 PES sessions. A session is a 10-minute stimulation, once per day. The sessions will be given on three consecutive days at optimal parameters, as reported by Fraser et al. (2003). During the second stimulation trial, the same method and same device will be used. However, the base-station will be set to 0 milliampere (mA), so Sham subjects do not receive any active electrical current.
  Interventions: Device: Pharyngeal Electrical Stimulation; Other: Sham treatment
- Sham treatment + Sham treatment in stroke patients (Sham Comparator): Max 8 patients will receive Sham twice. In the Sham condition, the same method and same device will be used. The time spent interacting with the patient will remain constant, including placement of the PES catheter which will be left in situ in the subject for the duration of intervention (10 minutes). However, the base-station will be set to 0 milliampere (mA), so Sham subjects do not receive any active electrical current.
  Interventions: Other: Sham treatment
- PES stimulation + PES stimulation in ICU patients (Experimental): Max 20 patients will receive PES stimulation twice. For patients, the protocol thus includes 2 stimulation trails. Each stimulation trial consists of 3 PES sessions, so they receive 6 PES sessions in total. A session is a 10-minute stimulation, once per day. The sessions will be given on three consecutive days at optimal parameters, as reported by Fraser et al. (2003).
  Interventions: Device: Pharyngeal Electrical Stimulation
- Sham treatment + Sham treatment in ICU patients (Experimental): Max 20 patients will receive Sham twice. In the Sham condition, the same method and same device will be used. The time spent interacting with the patient will remain constant, including placement of the PES catheter which will be left in situ in the subject for the duration of intervention (10 minutes). However, the base-station will be set to 0 milliampere (mA), so Sham subjects do not receive any active electrical current.
  Interventions: Other: Sham treatment

INTERVENTIONS:
Device: Pharyngeal Electrical Stimulation — A "Phagenyx" catheter is inserted trans-nasally. The catheter design incorporates a nasogastric feeding tube with built-in stimulation electrodes. The intervention consists of 3 PES sessions. A session is a 10-minute stimulation, once per day. The sessions will be given on three consecutive days at optimal parameters.
  Other Names: "Phagenyx"
  Arms: PES stimulation + PES stimulation in ICU patients; PES stimulation + PES stimulation in stroke patients; PES stimulation + Sham treatment in stroke patients; PES stimulation in volunteers
Other: Sham treatment — In the Sham condition, the same method and same device will be used. The time spent interacting with the patient will remain constant, including placement of the PES catheter which will be left in situ in the subject for the duration of intervention (10 minutes). However, the base-station will be set to 0 milliampere (mA), so Sham subjects do not receive any active electrical current.
  Other Names: Sham
  Arms: PES stimulation + Sham treatment in stroke patients; Sham treatment + Sham treatment in ICU patients; Sham treatment + Sham treatment in stroke patients; Sham treatment in volunteers

SUMMARY:
The goal of this clinical trial is to clarify which biomechanical aspects of swallowing are altered by Pharyngeal Electrical Stimulation (PES) in stroke patients, ICU patients and healthy volunteers.

The peripheral effect of PES intervention on the biomechanics of swallowing will be evaluated with High Resolution Manometry Impedance (HRMI).

DETAILED DESCRIPTION:
HRMI combines the evaluation of bolus flow patterns (impedance) and pressure (manometry) generated during swallowing.

20 healthy volunteers will participate, of which 10 will receive PES stimulation and 10 will receive Sham treatment.

Maximally 24 patients with dysphagia after acute stroke will be included. Group 1 will receive PES stimulation twice, group 2 will receive PES stimulation and afterwards Sham and group 3 will receive Sham twice.

Maximally 40 patients with Critical Illness Polyneuropathy/Myopathy or Post-Extubation Dysphagia will participate, of which 20 will receive PES stimulation and 20 will receive Sham treatment.

ELIGIBILITY:
Inclusion Criteria volunteers:

Healthy volunteers can participate in this study if they:

* Are aged between 18 and 80 years old
* Have no (history of) chronic disease/medication altering the gastrointestinal (GI) motility
* Have no (history of) gastric or gastrointestinal surgery (except appendectomy and cholecystectomy)
* Have no (history of) gastrointestinal disease or chronic GI symptoms (heartburn, indigestion/dyspepsia, bloating and constipation)
* Have FOIS score 7 or BEDQ score <10 at baseline
* Provide witnessed written informed consent prior to any study procedure And if they do not meet any of the exclusion criteria listed below.

Exclusion Criteria volunteers:

Healthy volunteers will be excluded if they:

* Are aged <18 years or >80 years
* Have (any history of) a chronic disease/medication altering the GI motility
* Have (any history of) gastric or gastrointestinal surgery (except appendectomy and cholecystectomy)
* Have (any history of) gastrointestinal disease or chronic GI symptoms (heartburn, indigestion/dyspepsia, bloating and constipation)
* Have a FOIS score <7 or a BEDQ score ≥ 10 at baseline
* Fail to provide witnessed written informed consent prior to any study procedure

Inclusion Criteria patients:

Dysphagic patients are eligible for study participation if they:

* Are admitted to the hospital because of acute stroke (acute means assessment within one month post stroke onset)

  * Hemorrhagic and ischemic stroke
  * Supratentorial and infratentorial stroke or have post-extubation dysphagia (PED) due to recent extubation following invasive mechanical ventilation (of any duration) by means of endotracheal tube or received (prolonged) intensive-care unit treatment leading to critical illness dysphagia due to (clinical suspicion of) critical illness polyneuropathy (CIP) and myopathy (CIM)
* Are aged between 18 and 85 years old
* Are medically stable, alert or arousable (Stroke: National Institutes of Health Stroke Scale (NIHSS) 0/1, ICU: Richmond Agitation-Sedation Scale (RASS) -1/0/+1 and Intensive Care Delirium Screening Checklist (ICDSC) <4)
* Have clinical (oropharyngeal) dysphagia well identified using the FOIS/DSRS/ BEDQ/PAS at baseline. In line with earlier studies(16,27), we use the following criteria: a DSRS score of 6 or higher; or a FOIS-score equal to or lower than 5; or a BEDQ score of 10 or higher or (when no oral food intake is possible and DSRS score is 12/FOIS score is 1) a PAS-score of 4 or higher
* Give (or have a witness to give) voluntary written informed consent And if they do not meet any of the exclusion criteria listed hereunder.

Exclusion Criteria patients:

Patients will be excluded from study participation if:

* They are aged <18 years or >85 years
* They have pre-existing neurogenic dysphagia or a condition that can cause dysphagia (e.g. advanced dementia, Parkinson's Disease, myasthenia gravis, motor neuron disease…);
* They have pre-existing non-neurogenic dysphagia (e.g. cancer, …);
* They have normal swallowing at baseline assessed with FOIS/DSRS/BEDQ/PAS
* When they participate in another interventional study, they must inform the researcher or study staff. They agree not to participate in another study simultaneously without having informed the researcher or study staff, and that participation may be refused for justified reasons.
* They receive or have received within one month prior to the intended PES treatment any form of non-invasive brain stimulation or percutaneous electrical stimulation therapy to treat dysphagia. (This is no issue, since this type of treatment is not performed at University Hospitals Leuven.)
* It is not possible to pass a standard nasogastric tube, for example, nasal, oral, pharyngeal or oesophageal anatomical abnormalities that preclude passage of a feeding tube, oral intubation, history of oesophageal perforation, stricture, pouch or resection, maxillofacial surgery, partial or total laryngectomy
* They have a cardiac or respiratory condition that might render the insertion of a catheter into the throat unsafe (Severe heart failure, end stage chronic obstructive pulmonary disease (COPD). Atrial fibrillation does not render the insertion of a catheter unsafe)
* They have a permanently implanted electrical device
* They are pregnant
* They present with an oropharyngeal infection. This should be treated and resolved before the PES catheter is inserted
* They require an MRI scan during PES treatment. Insertion of the PES catheter should either be delayed until such time as the MRI has been completed, or the PES catheter should be removed and discarded and a new catheter inserted after the MRI is completed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in pressure-flow metrics | Change from Baseline at 1-2 hours, 24-72 hours and one week (only in patients) after PES/Sham intervention.
  The primary outcome measure are alterations of the biomechanics of swallowing, assessed with HRMI. Analysis of these measurements results in pressure impedance metrics of deglutition, called Pressure Flow Analysis (PFA) parameters. These outcomes are numerical measures that can be compared to reference ranges to detect abnormality and to predict aspiration risk through derivation of a swallow risk index (SRI). An SRI > 15 indicates global swallowing dysfunction and aspiration risk, so higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Functional Oral Intake Scale | Change from Baseline at 24-72 hours and one week after last PES/Sham intervention
  The Functional Oral Intake Scale (FOIS) encompasses the amount and type of food that can be safely consumed, any special preparations of that food, any maneuvers or compensation being used to facilitate the swallow and the amount of supervision required if any. This valid, reliable, concise scale consists of seven levels that range from a patient who is unable to orally consume any food or liquid at Level 1, to a patient who is consuming an oral diet with no restrictions at Level 7. Higher scores mean a better outcome.
Brief Esophageal Dysphagia Questionnaire (BEDQ) | Change from Baseline at 24-72 hours and one week after last PES/Sham intervention
  The Brief Esophageal Dysphagia Questionnaire (BEDQ) is a 10-item self-report measure of oesophageal dysphagia symptom frequency (five items), severity (three items), and impaction (two items) with a total score ranging from 0 (asymptomatic) to 40. Higher scores indicate greater severity and frequency of oesophageal dysphagia symptoms, so a worse outcome.
Change in Dysphagia Severity Rating Scale (DSRS) in patients | Change from Baseline at 24-72 hours and one week after last PES/Sham intervention
  The Dysphagia Severity Rating Scale (DSRS) reflects the feeding status of patients across 3 domains: fluid modification, dietary adaptation and supervision requirements. The total score ranges from 0 (normal fluids, normal diet, and eating independently) to 12 (no oral fluids, no oral feeding). A higher score means a worse outcome.
Change in National Institutes of Health Stroke Scale (NIHSS) in stroke patients | Change from Baseline at 24-72 hours and one week after last PES/Sham intervention
  The National Institutes of Health Stroke Scale (NIHSS) is a reliable, valid 15-item impairment scale for measuring stroke severity. Item scores are summed to a total score ranging from 0 to 42 (the higher the score, the more severe the stroke: <5 limited stroke; 5-14 moderately severe stroke; 15-25 severe stroke; >25 very severe stroke). A higher score means a worse outcome.
Change in Penetration-Aspiration Scale (PAS) in patients | Change from Baseline at 24-72 hours and one week after last PES/Sham intervention
  The Penetration-Aspiration Scale (PAS) is an 8-point ordinal scale to describe penetration and aspiration events, primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled. Score 1 means that material does not enter the airway (no dysphagia). Score 8 means: material enters the airway, passes below the vocal folds and no effort is made to eject (severe dysphagia). A higher score means a worse outcome. These PAS scores are measured instrumentally by Fibreoptic Endoscopic Evaluation of Swallowing (FEES).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Rommel, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaam-Brabant, Belgium